CLINICAL TRIAL: NCT04719585
Title: Comparison of Opioid and Duloxetine for Postoperative Pain Control After Total Knee Arthroplasty: Randomized Controlled Trial
Brief Title: Comparison of Opioid and Duloxetine for Postoperative Pain Control After Total Knee Arthroplasty: RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Yong In, Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KC20MISI0531
Record Dates: First submitted 2021-01-06; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Total Knee Arthroplasty; Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Duloxetine group (Experimental): Prior to discharge, the drug is prescribed for a total of 6 weeks by dividing the duloxetine-administered group and the opioid-administering group, respectively. The administration period of duloxetine is 6 weeks. The follow-up periods for out-patient clinic are 2 weeks, 6 weeks, 3 months, 6 months, and 1 year after the TKA surgery. During the follow-up period, NSAIDs will be prescribed the same in both groups. As an additional rescue medication, 650 mg of acetaminophen will be allowed to use up to 2g per day.
  Interventions: Drug: Duloxetine vs. Opioid
- Active comparator: Opioid group (Active Comparator): Prior to discharge, the drug is prescribed for a total of 6 weeks by dividing the duloxetine-administered group and the opioid-administering group, respectively. The administration period of opioid is 6 weeks. The follow-up periods for out-patient clinic are 2 weeks, 6 weeks, 3 months, 6 months, and 1 year after the TKA surgery. During the follow-up period, NSAIDs will be prescribed the same in both groups. As an additional rescue medication, 650 mg of acetaminophen will be allowed to use up to 2g per day.
  Interventions: Drug: Duloxetine vs. Opioid

INTERVENTIONS:
Drug: Duloxetine vs. Opioid — Prior to discharge, the drug is prescribed for a total of 6 weeks by dividing the duloxetine-administered group and the opioid-administering group, respectively. The administration period of duloxetine or opioid is 6 weeks. The follow-up periods for out-patient clinic are 2 weeks, 6 weeks, 3 months, 6 months, and 1 year after the TKA surgery. During the follow-up period, NSAIDs will be prescribed the same in both groups. As an additional rescue medication, 650 mg of acetaminophen will be allowed to use up to 2g per day.

SUMMARY:
Serotonin-Norepinephrine Reuptake Inhibitor (SNRI) has recently been reported to be effective in controlling pain in persistent chronic pain caused by joint surgery and arthritis. However, opioids are important drugs that still play a pivotal role in pain control after surgery. In this study, we want to investigate the difference of the result among patients who undego total knee arthroplasty (TKA), of the result of pain control after TKA from SNRI administration of duloxetine and opioid in two groups. We designed a randomized controlled study (RCT) for the effect of post-TKA pain control to determine whether SNRI is effective in controlling post-TKA pain compared to Opioid, and whether there is a difference in side effects.

DETAILED DESCRIPTION:
For patients undergoing TKA for osteoarthritis of the knee joint, pain control will be performed using the same pain control technique (pain control using NSAID) until discharge (1 week after surgery) after surgery. By evaluating the Visual Analogue Scale (VAS), which is known as the patient's pain criterion, the study will be conducted only on patients whose score is more severe than 4 points. Among these subjects, only patients who agreed to the study will be assigned to the group taking duloxetine and the group taking opioids with the same probability according to the randomization table for one week after surgery, that is, upon discharge. In our hospital, almost all patients with total knee arthroplasty are discharged one week after surgery, except for special cases such as morbidity of systemic diseases such as cardiopulmonary dysfunction or acute infection after surgery.

Among the co-researchers, one researcher who is in charge of only patient assignment is selected, and the person in charge creates a randomization table through computer generated randomization. During the assignment process, the assignee will not know in advance the next assignment group, and the randomization table is kept in secret. The assignee does not intervene in any other process of this study, and participates only in the task of selecting the assigned group using random checks. The evaluation is evaluated by an evaluator who is not aware of the patient allocation according to the randomization table among researchers participating in the clinical study. Such a study plan will be fully explained to the patient in the process of seeking consent for the study before discharge, as it is recorded in detail in the subject description, and only patients who have obtained this consent will be the subject of the study.

This criterion is established because both duloxetine and opioid are not used for all patients after surgery, but for additional pain control after surgery. Prior to discharge, the drug is prescribed for a total of 6 weeks by dividing the duloxetine-administered group and the opioid-administering group, respectively. In general, if duloxetine is not taken for more than 10 weeks, the frequency of discontinuation syndrome that can occur after discontinuation is remarkably low, so the administration period of 6 weeks was set as the administration period. The follow-up periods for out-patient clinic are 2 weeks, 6 weeks, 3 months, 6 months, and 1 year after the TKA surgery. During the follow-up period, NSAIDs will be prescribed the same in both groups.

As an additional rescue medication, 650 mg of acetaminophen will be allowed to use up to 2g per day.

Before surgery, 1 week after surgery, 2 weeks, 6 weeks, 3 months, 6 months, 1 year The degree of pain will be measured using the VAS pain scale, WOMAC pain scale, Brief pain inventory (BPI), Intermittent and Constant Osteoarthritis The pain (ICOAP) score is used to measure additional pain scales in various ways. In addition, SF-36 will be measured before surgery, at 6 weeks, 3 months, 6 months, and 1 year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults over age 19
* Patients undergoing total knee arthroplasty for osteoarthritis of the knee joint
* Patients with a pain VAS scale of 4 or more out of 10 after TKA with a pain in the knee joint during daily activities on flat ground
* Patients who are willing or able to follow doctor's instructions, including joint exercises
* Patients not participating in other clinical trials
* Patients who have received sufficient explanation for this clinical trial and agreed to participate

Exclusion Criteria:

* Patients with secondary knee osteoarthritis
* Patients with hypersensitivity reactions and serious side effects to duloxetine or opioid
* Patients with inflammatory arthritis or crystalline arthritis
* Local infection to the lower extremities of the pain area, sepsis, or previous neurological abnormalities.
* Patients who underwent meniscus surgery on the knee joint in the painful area
* If there is construction or deformation of the knee joint in the pain area
* Patients with serious heart-related diseases such as cardiac arrest, a history of cerebral infarction, or ischemic heart disease
* Patients with high blood pressure with poor blood pressure control (Systolic Blood Pressure of> 150 mmHg or Diastolic Blood Pressure> 95 mmHg)
* Patients with abnormal liver function (ALT)> 2.0 times the upper limit of normal (ULN) or blood urea nitrogen (BUN) or serum creatinine> 2.0 times ULN)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Pain Visual Analogue Scale | changes of the VAS score from the day before TKA operation and at postoperative 1, 2, 6, 12, 24th weeks and 1 year
  score ranges 0 to 10, higher score means more painful
Brief pain inventory (BPI) | changes of the BPI score from the day before TKA operation and at postoperative 1, 2, 6, 12, 24th weeks and 1 year
  includes 7 categories. each category score ranges 0 to 10, higher score means more painful

SECONDARY OUTCOMES:
WOMAC(Western Ontario and McMaster University Arthritis Index ) pain scale | changes of the WOMAC score from the day before TKA operation and at postoperative 1, 2, 6, 12, 24tn weeks and 1 year
  The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). higher score means more painful.
Intermittent and Constant Osteoarthritis pain (ICOAP) score | changes of the ICOAP score from the day before TKA operation and at postoperative 1, 2, 6, 12, 24tn weeks and 1 year
  11-item tool that assess pain at knee joint. The 11 items are scored froma 0 to 4 with 0 being no pain and 4 being extreme pain
SF-36(Short Form Health Survey - 36) score | changes of the SF-36 score from the day before TKA operation and at postoperative 1, 2, 6, 12, 24tn weeks and 1 year
  a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability
Range of Motion | The day before TKA operation, postoperative 1, 2, 6, 12, 24 weeks and 1 year

IPD SHARING:
Plan to Share IPD: No